CLINICAL TRIAL: NCT01894373
Title: Autologous Cytokine Induced Killer Cells as Adjuvant Adoptive Immunotherapy in Patients With Psoriasis
Brief Title: Autologous Cytokine Induced Killer Cells (CIK) for Patients With Severe Psoriasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Ph.D, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HWD301
Record Dates: First submitted 2013-06-27; First posted 2013-07-10 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2015-06

CONDITIONS: Psoriasis; Adoptive Immunotherapy
MeSH Terms: conditions — Psoriasis | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CIK, psoriasis (Experimental)
  Interventions: Drug: Adoptive Immunotherapy; Biological: CIK

INTERVENTIONS:
Drug: Adoptive Immunotherapy — Biological: in vitro expanded Cytokine Induced Killer (CIK) cells Procedure: Infusion of autologous CIK cells
Biological: CIK

SUMMARY:
to determine the therapeutic roles of CIK cells on patients with psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Have ever had a physician's diagnosis of chronic moderate to severe plaque psoriasis and be a candidate for treatment with CIK Are being treated with or initiating CIK therapy at the time of enrollment Be able to provide written informed consent Be willing and able to fully to participate for the duration of patient follow-up (5 years)

Exclusion Criteria:

* PUVA or Grenz ray therapy within 4 weeks prior to randomisation. UVB therapy within 2 weeks prior to randomisation. Systemic treatment with biological therapies (marketed or otherwise) with a possible effect on psoriasis (e.g., alefacept, efalizumab, etanercept, infliximab) within 3 months prior to randomisation.

Systemic treatment other than biologicals with a possible effect on psoriasis (e.g., corticosteroids, vitamin D analogues, retinoids, hydroxycarbamide, azathioprine, meth-otrexate, cyclosporine, other immunosuppressants) within 4 weeks prior to randomisation.

Any topical treatment of the scalp (except for medicated shampoos and emollients) within 2 weeks prior to randomisation (medicated shampoos/emollients are not allowed during the double-blind phase). Shampoos containing corticosteroids, e.g. Clobex®, are not allowed within 2 weeks prior to randomisation.

Planned use of topical treatment for psoriasis of the trunk or limbs, besides study medication, during the study with the exceptions of: • emollient • medications used to treat psoriasis of the skin folds and/or genitals (any medication may be used for this purpose apart from Class 1-5 corticosteroids.

Topical treatment of the face with Class 1-5 corticosteroids within 2 weeks prior to randomisation.

Planned initiation of, or changes to, concomitant medication that could affect psoriasis (e.g., beta blockers, anti-malaria drugs, lithium) during the double-blind phase of the study.

Treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within 4 weeks prior to randomisation.

Planned use of chemical treatments of the hair (eg relaxers, 'perms', or colourings) during the double-blind phase of the study.

Current diagnosis of erythrodermic, exfoliative or pustular psoriasis. Patients with any of the following conditions also present on psoriatic areas of the scalp or trunk/limbs: viral (e.g. herpes or varicella) lesions of the skin, fungal or bacterial skin infections, parasitic infections, skin manifestations in relation to tuberculosis or syphilis, rosacea, acne rosacea, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, ulcers or wounds.

Other inflammatory skin diseases that may confound the evaluation of psoriasis of the scalp or trunk/limbs.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
therapeutic roles of CIK on psoriasis | 1 year
  changes of area and extent of skin lesions

SECONDARY OUTCOMES:
Occurrence of study related adverse events | within 2 weeks
  adverse effect after CIK cell infusion

OTHER OUTCOMES:
infiltration of immune cells under skin | 6 months
  aberrant infiltration of immune cells within the full-thickness of skin by skin biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Han weidong, doctor, Study Director — Institute of immunology，Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Dai H, Zhou Y, Tong C, Guo Y, Shi F, Wang Y, Shen P. Restoration of CD3+CD56+ cell level improves skin lesions in severe psoriasis: A pilot clinical study of adoptive immunotherapy for patients with psoriasis using autologous cytokine-induced killer cells. Cytotherapy. 2018 Sep;20(9):1155-1163. doi: 10.1016/j.jcyt.2018.07.003. Epub 2018 Aug 9. PMID 30100374